CLINICAL TRIAL: NCT03834818
Title: COMPAS Trial. Collecting Outcomes and Managing Pain After Surgery: Predicting Patients at High Risk for Chronic Opioid Use and Creating Algorithms to Responsibly Tailor Opioid Prescribing and Weaning After Surgery
Brief Title: Collecting Outcomes and Managing Pain After Surgery
Acronym: COMPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00094157
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Surgery
Keywords: opioid use; pain; surgery; orthopedic surgery; orthopedic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Patients undergoing orthopedic surgery at Duke Health will be eligible for enrollment. Additionally, all potential participants must be an adult at least 18 years of age, speak and read English, own a smartphone they are willing to use for the study, and live in the United States of America. All study assessments will take place on the app and other than baseline screening all assessments will take place after surgery until the patient stops taking opioids. Patients will be approached in the orthopedic clinic up to the day of surgery and asked if they are willing to be screened for inclusion. If they accept the screening request a link will be emailed to them or a QR code supplied that permits them to download the study app on their phone. Screening, consent, and all study data collection will occur from the app launch. All data will be collected after enrollment and consent through the Medable Research Application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMPAS Participants (Experimental): Patents between the ages of 18 and 90 who are undergoing orthopedic surgery at Duke Health will be eligible for enrollment.
  Interventions: Behavioral: COMPAS Participants

INTERVENTIONS:
Behavioral: COMPAS Participants — The schedule of events for this study are as follows:
  Day 1 Pre-Surgery:
  * Download the Medable App
  * Register to the study
  * Validated Questionnaires
  * Active Task
  Every Day
  * 9:00 a.m. Daily Questions
  * 9:00 p.m. Daily Questions
  Outcome Surveys and Active Task:
  * Day 1 Pre-Surgery
  * 1-Week Post Operation
  * 2-Weeks Post Operation
  * 1-Month Post Operation
  * 3-Months Post Operation
  * 6-Months Post Operation

SUMMARY:
The primary aim of this study is to measure pain and psychosocial patient reported outcomes, objective functionality, and actual daily at home opioid usage in orthopedic patients. The study's goal following the data collection is to predict which patients are at high risk for chronic opioid use.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-90 years old who are undergoing elective orthopedic surgery at Duke Health.
* Patients must have their own smartphone IOS or Android device.
* Patients must be able to read English.

Exclusion Criteria:

* Lacking capacity to provide consent.
* Cannot read English
* Under 18 years of age
* Older than 90 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Reported Pain of Participants measured via PROMIS-29 | 6 Months
  28 Questions regarding pain are ranked on a 5-point Likert Scale with 1 meaning "not at all" and 5 meaning "very much".
Reported Pain of Participants measured via PROMIS-29 | 6 Months
  One question on an 11-point rating scale for pain intensity, with 0 meaning "no pain" and 10 meaning "worst imaginable pain".
Reported Pain of Participants measured via Pain Catastrophizing pain scale. | 6 Months
  Statements regarding pain are rated on a scale from 0 to 4 with 0 meaning "not at all" and 4 meaning "all the time"
Opioid Use of Participants | 6 months
  Total number of patients with self reported use of opioids.
Practicality of Mobile Application | 6 Months
  How long participants actively use the app to track their opined use and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bullock, MD, Principal Investigator — Duke University
Locations (1):
- Duke Orthopaedics, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No